CLINICAL TRIAL: NCT01114139
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Trial of Ferumoxytol for the Treatment of Iron Deficiency Anemia
Brief Title: A Trial Comparing Ferumoxytol With Placebo for the Treatment of Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMAG-FER-IDA-301
Record Dates: First submitted 2010-04-29; First posted 2010-04-30 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency anemia; Feraheme; ferumoxytol; IDA
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferumoxytol (Experimental): Participants received a total of 2 doses of IV ferumoxytol 510 milligrams (mg) (17 milliliters [mL]). The first IV 510 mg dose was administered on Day 1 (Baseline) and second dose 2 to 8 (5±3) days after the first dose, for a total cumulative dose of 1.02 grams (g).
  Interventions: Drug: Ferumoxytol
- Placebo (Placebo Comparator): Participants received a total of 2 doses of IV saline (17 mL). The first IV dose was administered on Day 1 (Baseline) and second dose 2 to 8 (5±3) days after the first dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ferumoxytol — IV Ferumoxytol
  Other Names: Feraheme
  Arms: Ferumoxytol
Other: Placebo — IV Placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of intravenous (IV) ferumoxytol compared with placebo for the treatment of iron deficiency anemia (IDA).

DETAILED DESCRIPTION:
This Phase III, randomized, double-blind, placebo-controlled, multicenter clinical study evaluated the safety and efficacy of ferumoxytol compared with placebo for the treatment of IDA, specifically in adult patients with IDA who have a history of unsatisfactory oral iron therapy or in whom oral iron could not be used. The effect of ferumoxytol on hemoglobin, iron parameters and patient reported outcomes (PROs) compared with placebo was evaluated. Investigators were blinded to key laboratory parameters that could potentially unblind the treatment arms of the study, eg, hemoglobin [Hgb], hematocrit [Hct], iron, ferritin, total iron binding capacity [TIBC], and transferrin saturation [TSAT], and neither the Investigators nor the subjects were aware of their treatment assignment, hemoglobin or other laboratory values.

ELIGIBILITY:
Key Inclusion Criteria include:

1. Males and females ≥18 years of age
2. Participants with IDA defined as having:

   1. Hemoglobin <10.0 g/deciliter (dL)
   2. Transferrin saturation <20%
3. Participants who have a history of unsatisfactory oral iron therapy or in whom oral iron cannot be used
4. Female participants of childbearing potential who are sexually active must be on an effective method of birth control for at least 1 month prior to screening and agree to remain on birth control until completion of participation in the study

Key Exclusion Criteria include:

1. History of allergy to IV iron
2. Allergy to two or more classes of drugs
3. Participants on dialysis or with an estimated glomerular filtration rate <30 mL/minute/1.73 m^2
4. Female participants who are pregnant, intend to become pregnant, are breastfeeding, within 2 weeks postpartum, or have a positive serum/urine pregnancy test
5. Hemoglobin ≤7.0 g/dL
6. Serum ferritin >600 nanograms/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2010-06-19 (Actual); Primary Completion 2012-02-27 (Actual); Study Completion 2012-10-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (144):
- United States (108):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, Mobile, Alabama
  - Clinical Trial Site, Montgomery, Alabama
  - Clinical Trial Site, Green Valley, Arizona
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Tucson, Arizona
  - Clinical Trial Site, Alhambra, California
  - Clinical Trial Site, Anaheim, California
  - Clinical Trial Site, Bakersfield, California
  - Clinical Trial Site, Buena Park, California
  - Clinical Trial Site, Colton, California
  - Clinical Trial Site, Fresno, California
  - Clinical Trial Site, Glendale, California
  - Clinical Trial Site, Laguna Hills, California
  - Clinical Trial Site, Lakewood, California
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Mission Hills, California
  - Clinical Trial Site, Orange, California
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, Pueblo, Colorado
  - Clinical Trial Site, Bristol, Connecticut
  - Clinical Trial Site, Groton, Connecticut
  - Clinical Trial Site, Newark, Delaware
  - Clinical Trial Site, Boynton Beach, Florida
  - Clinical Trial Site, Clearwater, Florida
  - Clinical Trial Site, Hialeah, Florida
  - Clinical Trial Site, Holiday, Florida
  - Clinical Trial Site, Inverness, Florida
  - Clinical Trial Site, Margate, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Miami Lakes, Florida
  - Clinical Trial Site, Naples, Florida
  - Clinical Trial Site, Ocala, Florida
  - Clinical Trial Site, Vero Beach, Florida
  - Clinical Trial Site, Wellington, Florida
  - Clinical Trial Site, West Palm Beach, Florida
  - Clinical Trial Site, Winter Park, Florida
  - Clinical Trial Site, Zephyrhills, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Columbus, Georgia
  - Clinical Trial Site, Decatur, Georgia
  - Clinical Trial Site, Dublin, Georgia
  - Clinical Trial Site, Rome, Georgia
  - Clinical Trial Site, Sandy Springs, Georgia
  - Clinical Trial Site, Savannah, Georgia
  - Clinical Trial Site, Stockbridge, Georgia
  - Clinical Trial Site, Aurora, Illinois
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Evergreen Park, Illinois
  - Clinical Trial Site, Skokie, Illinois
  - Clinical Trial Site, Springfield, Illinois
  - Clinical Trial Site, Indianapolis, Indiana
  - Clinical Trial Site, Wichita, Kansas
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Bethesda, Maryland
  - Clinical Trial Site, Hollywood, Maryland
  - Clinical Trial Site, Prince Frederick, Maryland
  - AMAG Pharmaceuticals, Inc., Waltham, Massachusetts
  - Clinical Trial Site, Bay City, Michigan
  - Clinical Trial Site, Saginaw, Michigan
  - Clinical Trial Site, Wyoming, Michigan
  - Clinical Trial Site, Kansas City, Missouri
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, Lawrenceville, New Jersey
  - Clinical Trial Site, Neptune City, New Jersey
  - Clinical Trial Site, Plainsboro, New Jersey
  - Clinical Trial Site, Somerville, New Jersey
  - Clinical Trial Site, Voorhees Township, New Jersey
  - Clinical Trial Site, Albuquerque, New Mexico
  - Clinical Trial Site, Brooklyn, New York
  - Clinical Trial Site, Goshen, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Raleigh, North Carolina
  - Clinical Trial Site, Wilmington, North Carolina
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Bismarck, North Dakota
  - Clinical Trial Site, Akron, Ohio
  - Clinical Trial Site, Beavercreek, Ohio
  - Clinical Trial Site, Canton, Ohio
  - Clinical Trial Site, Carlisle, Ohio
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Dayton, Ohio
  - Clinical Trial Site, Marion, Ohio
  - Clinical Trial Site, Mentor, Ohio
  - Clinical Trial Site, Middletown, Ohio
  - Clinical Trial Site, Zanesville, Ohio
  - Clinical Trial Site, Norman, Oklahoma
  - Clinical Trial Site, Jenkintown, Pennsylvania
  - Clinical Trial Site, Levittown, Pennsylvania
  - Clinical Trial Site, East Providence, Rhode Island
  - Clinical Trial Site, Columbia, South Carolina
  - Clinical Trial Site, Greer, South Carolina
  - Clinical Trial Site, Myrtle Beach, South Carolina
  - Clinical Trial Site, North Charleston, South Carolina
  - Clinical Trial Site, Orangeburg, South Carolina
  - Clinical Trial Site, Rapid City, South Dakota
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Arlington, Texas
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Laredo, Texas
  - Clinical Trial Site, Longview, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Spring, Texas
  - Clinical Trial Site, Orem, Utah
  - Clinical Trial Site, Chesapeake, Virginia
  - Clinical Trial Site, Norfolk, Virginia
- Canada (7):
  - Clinical Trial Site, Vancouver, British Columbia
  - Clinical Trial Site, Saint John, New Brunswick
  - Clinical Trial Site, London, Ontario
  - Clinical Trial Site, Scarborough Village, Ontario
  - Clinical Trial Site, Thornhill, Ontario
  - Clinical Trial Site, Vaughan, Ontario
  - Clinical Trial Site, Pointe-Claire, Quebec
- Hungary (5):
  - Clinical Trial Site, Békéscsaba
  - Clinical Trial Site, Gyula
  - Clinical Trial Site, Komárom
  - Clinical Trial Site, Szekszárd
  - Clinical Trial Site, Vác
- India (15):
  - Clinical Trial Site, Hyderabad, Andhra Pradesh
  - Clinical Trial Site, Secunderabad, Andhra Pradesh
  - Clinical Trial Site, Visakhapatnam, Andhrapradesh
  - Clinical Trial Site, Guwahati, Assam
  - Clinical Trial Site, Bangalore, Karnataka
  - Clinical Trial Site, Mangalore, Karnataka
  - Clinical Trial Site, Aurangabad, Maharashtra
  - Clinical Trial Site, Nagpur, Maharashtra
  - Clinical Trial Site, Nashik, Maharashtra
  - Clinical Trial Site, Pune, Maharashtra
  - Clinical Trial Site, Jaipur, Rajasthan
  - Clinical Trial Site, Chennai, Tamil Nadu
  - Clinical Trial Site, Coimbatore, Tamil Nadu
  - Clinical Trial Site, Madurai, Tamil Nadu
  - Clinical Trial Site, Lucknow, Uttar Pradesh
- Latvia (4):
  - Clinical Trial Site, Daugavpils
  - Clinical Trial Site, Riga
  - Clinical Trial Site, Valmiera
  - Clinical Trial Site, Ventspils
- Poland (5):
  - Clinical Trial Site, Bialystok
  - Clinical Trial Site, Sopot
  - Clinical Trial Site, Warsaw
  - Clinical Trial Site, Wroclaw
  - Clinical Trial Site, Zgierz

REFERENCES:
- [Background] Vadhan-Raj S, Strauss W, Ford D, Bernard K, Boccia R, Li J, Allen LF. Efficacy and safety of IV ferumoxytol for adults with iron deficiency anemia previously unresponsive to or unable to tolerate oral iron. Am J Hematol. 2014 Jan;89(1):7-12. doi: 10.1002/ajh.23582. Epub 2013 Sep 30. PMID 23983177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to enrollment for adult participants with iron deficiency anemia (IDA), defined as hemoglobin <10.0 gram (g)/deciliter (dL) and transferrin saturation (TSAT) <20%, and a history of unsatisfactory oral iron therapy or in whom oral iron could not be used.
Groups:
- Ferumoxytol: Participants received a total of 2 doses of intravenous (IV) ferumoxytol 510 milligrams (mg) (17 milliliters [mL]). The first IV 510 mg dose was administered on Day 1 (Baseline) and second dose 2 to 8 (5±3) days after the first dose, for a total cumulative dose of 1.02 g.
Period: Overall Study
Arm/Group | Ferumoxytol | Placebo
Started | 609 | 203
Received at Least 1 Dose of Study Drug | 608 | 200
Completed (Completed is defined as had study drug and Week 5 visit.) | 569 | 187
Not Completed | 40 | 16
Not completed — Adverse Event | 3 | 2
Not completed — Lost to Follow-up | 15 | 3
Not completed — Withdrawal by Subject | 17 | 6
Not completed — Other-Missed 1 visit | 1 | 0
Not completed — Other-Protocol Violation | 1 | 0
Not completed — Other-Out of window for study drug dose | 1 | 0
Not completed — Other-Participant falsified records | 0 | 1
Not completed — Other-Participant went on hospice | 0 | 1
Not completed — Other-Physician changed treatment | 1 | 0
Not completed — Other-Withdrew prior to receiving dose | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) Population: Any randomized participant who had any exposure to study drug (ferumoxytol or placebo) and was based upon randomized treatment assignment.
Groups:
- Ferumoxytol: Participants received a total of 2 doses of IV ferumoxytol 510 mg (17 mL). The first IV 510 mg dose was administered on Day 1 (Baseline) and second dose 2 to 8 (5±3) days after the first dose, for a total cumulative dose of 1.02 g.
- Total: Total of all reporting groups
Arm/Group | Ferumoxytol | Placebo | Total
Number analyzed (Participants) | 608 | 200 | 808
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (13.82) | 46.0 (13.58) | 45.1 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 542 | 178 | 720
  Male | 66 | 22 | 88

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Achieved A ≥2.0 g/dL Increase In Hemoglobin At Any Time From Baseline To Week 5
Description: Participants who achieved a ≥2.0 g/dL increase in hemoglobin at any time from Baseline up to Week 5 are presented. Increase in hemoglobin at any time from Baseline up to Week 5 was calculated for each participant based on:
  Hemoglobin Change = Hemoglobin (Week X) - Hemoglobin (Baseline), where Week X was any post-Baseline visit up to and including Week 5.
  Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. Participants with no post-Baseline hemoglobin values were classified as not achieving a ≥2.0 g/dL increase.
  Statistical analysis was performed for data up to Week 5 only.
Time Frame: Baseline (Day 1) through Week 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Ferumoxytol | Placebo
Number analyzed (Participants) | 608 | 200
Participants
  Up to Week 2 | 252 | 5
  Up to Week 3 | 386 | 7
  Up to Week 4 | 460 | 8
  Up to Week 5 | 493 | 11
Statistical Analysis 1: Comparison: Ferumoxytol vs Placebo; Participants who achieved a ≥2.0 g/dL increase in hemoglobin from Baseline up to Week 5 were analyzed. Statistical comparison was performed for data up to Week 5 only. Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information; Test type: Superiority — The 95% confidence interval was calculated using the large sample assumption; p < 0.0001, Cochran-Mantel-Haenszel; The p-value is the result of the Cochran-Mantel-Haenszel test, adjusted for Baseline hemoglobin level and underlying condition; Treatment Difference = 75.59, 95% CI 2-sided [71.15 to 80.02] — The treatment difference (ferumoxytol - placebo) was expressed as a percentage

2. Secondary Outcome: Mean Change In Hemoglobin From Baseline To Week 5
Description: Mean change in hemoglobin from Baseline to Week 5 was calculated for each participant as:
  Hemoglobin Change = Hemoglobin (Week X) - Hemoglobin (Baseline), where Week X was any post-Baseline visit up to and including Week 5. Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. If the Week 5 hemoglobin value was missing, the change from Baseline was imputed to be zero. Participants without any post-Baseline hemoglobin values were treated as non-responders.
Time Frame: Baseline (Day 1), Week 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferumoxytol | Placebo
Number analyzed (Participants) | 608 | 200
g/dL | 2.6 (1.52) | 0.1 (0.89)

3. Secondary Outcome: Participants Achieving A Hemoglobin Level ≥12.0 g/dL At Any Time From Baseline To Week 5
Description: Participants who achieved a ≥12.0 g/dL hemoglobin level at any time from Baseline up to Week 5 are presented. Increase in hemoglobin at any time from Baseline up to Week 5 was calculated for each participant based on:
  Hemoglobin Change = Hemoglobin (Week X) - Hemoglobin (Baseline), where Week X was any post-Baseline visit up to and including Week 5. Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. Participants without any post-Baseline hemoglobin values were treated as non-responders.
Time Frame: Baseline (Day 1) through Week 5
Population: ITT Population: Any randomized participant who had any exposure to study drug (ferumoxytol or placebo) and was based upon randomized treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ferumoxytol | Placebo
Number analyzed (Participants) | 608 | 200
Participants
  Up to Week 2 | 33 | 3
  Up to Week 3 | 131 | 5
  Up to Week 4 | 240 | 5
  Up to Week 5 | 307 | 6

4. Secondary Outcome: Mean Change In TSAT From Baseline To Week 5
Description: Mean change in TSAT from Baseline to Week 5 was calculated for each participant as: TSAT Change = TSAT (Week 5) - TSAT (Baseline).
  TSAT, measured as a percentage, was part of the iron panel laboratory evaluations. Of the transferrin available to bind iron, this value indicates how much serum iron is bound. For example, a value of 20% means that 20% of iron-binding sites of transferrin are being occupied by iron. Baseline was defined as the Day 1 value (prior to injection of study drug). The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. If the Week 5 TSAT value was missing, the change from Baseline was imputed to be zero.
Time Frame: Baseline (Day 1), Week 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Ferumoxytol | Placebo
Number analyzed (Participants) | 608 | 200
percentage of saturation | 11.4 (15.06) | 0.4 (5.81)

5. Secondary Outcome: Mean Change In Functional Assessment Of Chronic Illness Therapy (FACIT)-Fatigue Score From Baseline To Week 5
Description: The FACIT-Fatigue questionnaire is a 13-item questionnaire designed and validated to specifically assess the presence and impact of treatment on fatigue and related symptoms, such as tiredness, on health-related quality of life in anemic participants with cancer. The questionnaire has 13 items, each measured on a 4-point Likert scale. Scoring ranges from 0 (the most fatigued) to 52 (the least fatigued) points, with higher scores representing better functioning or less fatigue.
  Mean change in FACIT-Fatigue Score from Baseline to Week 5 was calculated for each participant as:
  FACIT-Fatigue Score Change = FACIT-Fatigue Score (Week 5) - FACIT-Fatigue Score (Baseline).
  Baseline was defined as the Day 1 value (prior to first dose of study drug).The screening or most recent value prior to Day 1 was used for any participant with missing Day 1 information. If the Week 5 FACIT-Fatigue Score value was missing, the change from Baseline was imputed to be zero.
Time Frame: Baseline (Day 1), Week 5
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ferumoxytol | Placebo
Number analyzed (Participants) | 608 | 200
units on a scale | 11.7 (11.73) | 6.8 (9.51)

6. Secondary Outcome: Time To Hemoglobin Increase Of ≥2.0 g/dL Or A Hemoglobin Value Of ≥12.0 g/dL From Baseline
Description: The time to hemoglobin increase of ≥2.0 g/dL or hemoglobin value of ≥12.0 g/dL was defined as the days from Baseline (Day 1) to the first time the participant had an increase in hemoglobin of ≥2.0 g/dL or hemoglobin value of ≥12.0 g/dL, and was calculated using a Kaplan-Meier curve. Participants who did not have a hemoglobin increase of ≥2.0 g/dL or to a hemoglobin level ≥12.0 g/dL were censored at their last visit day. Participants without any post-Baseline study visits were not included.
Time Frame: From Baseline (Day 1) up to Week 5
Population: as for baseline characteristics
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | Ferumoxytol | Placebo
Number analyzed (Participants) | 608 | 200
Days | 23.5 [15.0 to 29.0] | 42.5 [44 to NA] — Insufficient number of participants with events.

ADVERSE EVENTS:
Arm/Group | Ferumoxytol | Placebo
Serious Adverse Events (participants affected / at risk) | 16/608 | 6/200
Other Adverse Events (participants affected / at risk) | 198/608 | 56/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ferumoxytol (N=608) | Placebo (N=200)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Disease Progression (General disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0/542 | 1/178
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferumoxytol (N=608) | Placebo (N=200)
Abdominal Pain (Gastrointestinal disorders) | 11 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 1
Constipation (Gastrointestinal disorders) | 10 | 3
Diarrhoea (Gastrointestinal disorders) | 17 | 6
Nausea (Gastrointestinal disorders) | 28 | 5
Toothache (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 12 | 2
Fatigue (General disorders) | 12 | 3
Oedema Peripheral (General disorders) | 10 | 1
Pyrexia (General disorders) | 7 | 1
Nasopharyngitis (Infections and infestations) | 16 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 2
Urinary Tract Infection (Infections and infestations) | 17 | 6
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 7 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 1
Dizziness (Nervous system disorders) | 24 | 7
Dysgeusia (Nervous system disorders) | 9 | 1
Headache (Nervous system disorders) | 35 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 12 | 0
Hypertension (Vascular disorders) | 9 | 0
Hypotension (Vascular disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no multi-site publication within 18 months after Study has been completed or terminated at all Study sites, and all data have been received by Sponsor, Site, and Site Management Organization (SMO) shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 180 days to allow Sponsor to protect its interests.